CLINICAL TRIAL: NCT06528171
Title: Specific Markers of Covid-long Syndrome: Identifying the Mechanisms Involved With a View to Defining Diagnostic Criteria
Brief Title: Covid-19 Long Immunité IMagerie (CLIIM)
Acronym: CLIIM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 23-RECHMIE-01
Record Dates: First submitted 2024-07-29; First posted 2024-07-30 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: COVID Long-Haul
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Covid-long (CL+) (Other): Assessment of musculoskeletal disorders, cognitive and neurocognitive assessments, Behavioral assessment, Work Difficulty Scale, Digital testing, brain MRI, Biological Analysis
  Interventions: Procedure: Brain MRI; Biological: Specific blood samples
- Acute Covid (CL-) (Other): Brain MRI, Biological Analysis
  Interventions: Procedure: Brain MRI; Biological: Specific blood samples

INTERVENTIONS:
Procedure: Brain MRI — non injected brain MRI
Biological: Specific blood samples — blood samples to find immunological and inflammatory markers

SUMMARY:
Covid-long pathology affects a large number of patients, and represents a major medical, economic and societal challenge. To date, we have no objective criterion for a definitive diagnosis, nor any predictive tool for monitoring the evolution of Covid-long. Based on recruitment from the infectious diseases department of Nice University Hospital, the investigator's team wants to conduct an innovative pathophysiological study to better define the disease and identify specific biomarkers that could subsequently be used as a diagnostic tool for Covid-long. 120 participants will be initially included for the model learning phase: 60 controls in the CL- cohort and 60 patients in the CL+ cohort. Then 80 patients (40 CL+ and 40 Cl-) will be enrolled for the model validation phase.

ELIGIBILITY:
FOR CL+ PATIENTS

Inclusion Criteria:

* Case definition in line with WHO Delphi process

Exclusion Criteria:

* History of chronic fatigue syndrome diagnosed before or after Covid.
* History of progressive psychiatric pathology.
* History of acute Covid requiring admission to intensive care and mechanical ventilation.
* No social security affiliation.

FOR CONTROL (CL-)

Inclusion Criteria:

* History of acute COVID-19, mild, moderate or severe (episode at least 3 months at the time of inclusion).
* Absence of persistent symptoms more than 3 months after first Covid symptoms (or mild not affecting daily activities).

Exclusion Criteria:

* History of progressive psychiatric pathology.
* History of acute Covid requiring admission to intensive care and mechanical ventilation.
* No social security affiliation.
* Pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-12-06 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Predictive model of Covid-long | 24 months
  Build and validate a multivariate predictive model of Covid-long considering immunological, inflammatory and brain imaging markers.

SECONDARY OUTCOMES:
Evolution of these markers over time | 24 months
  Comparison of data over time between cohorts (CL+ vs. CL-)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de NICE, Nice, France

IPD SHARING:
Plan to Share IPD: No
Not planned